CLINICAL TRIAL: NCT04741607
Title: Alveolar Ridge Preservation With Immediate or Late Implant Placement: a Multicenter Randomized Controlled Trial
Brief Title: Immediate Versus Late Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-08574
Record Dates: First submitted 2020-10-17; First posted 2021-02-05 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Esthetics
Keywords: connective tissue graft; dental implant, single tooth; immediate; ridge preservation

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled study with 2 treatment arms (control: delayed implant placement; test: immediate implant placement) and 6 centers
Who Masked: Investigator, Outcomes Assessor
Masking Description: As this RCT concerns a surgical intervention, patients and treating clinicians can not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Delayed implant placement
  Interventions: Device: Implant placement (BLX implant system, Straumann, Basel, Switzerland); Procedure: Ridge preservation (Bio-Oss Collagen 250 mg, Geistlich Pharma AG, Wolhusen, Switserland); Procedure: Socket seal (Mucograft Seal, Geistlich Pharma AG, Wolhusen, Switserland)
- Test group (Experimental): Immediate implant placement
  Interventions: Device: Implant placement (BLX implant system, Straumann, Basel, Switzerland); Procedure: Ridge preservation (Bio-Oss Collagen 250 mg, Geistlich Pharma AG, Wolhusen, Switserland)

INTERVENTIONS:
Device: Implant placement (BLX implant system, Straumann, Basel, Switzerland) — Implants are placed after a healing period of 4 months (delayed implant placement, control group) or immediately after tooth extraction and ridge preservation (immediate implant placement, test group).
Procedure: Ridge preservation (Bio-Oss Collagen 250 mg, Geistlich Pharma AG, Wolhusen, Switserland) — Ridge preservation is performed by inserting a collagen-enriched DBBM (Bio-Oss Collagen 250 mg, Geistlich Pharma AG, Wolhusen, Switserland) in the empty extraction socket (delayed implant placement, control group) or by filling the gap between the implant and buccal bone wall (immediate implant placement, test group).
Procedure: Socket seal (Mucograft Seal, Geistlich Pharma AG, Wolhusen, Switserland) — The occlusal aspect of the grafted socket in the delayed implant placement/control group is closed with a collagen matrix.
  Arms: Control group

SUMMARY:
Patients in need of a single implant in the premaxilla will be invited to participate in this multicenter randomized controlled trial (RCT). Prior to surgery, a small-field low-dose cone beam computed tomography (CBCT) is taken to verify the integrity of the facial bone wall and an adequate amount of apical and palatal bone dimensions. Sixty patients will be randomly allocated to the test group or control group in 6 centers. Each center receives 10 sealed envelopes (5 are internally labelled with 'delayed implant placement' and 5 with 'immediate implant placement').

For each patient a digital planning is performed in implant planning software and a tooth-supported surgical guide is fabricated prior to tooth extraction.

In the control group, alveolar ridge preservation is performed following tooth extraction. After a healing period of 4 months, a single implant is installed.

In the test group, a single implant is installed immediately after tooth extraction and ridge preservation is performed by filling the gap between the facial bone wall and the implant surface.

A provisional crown is placed at the day of implant surgery, which is replaced by a permanent one 3m later.

Six months after tooth extraction and subsequent ridge preservation, the need for soft tissue grafting is assessed on the base of predetermined criteria (primary outcome measure). Soft tissue augmentation is performed by inserting a palatal connective tissue graft (CTG) into the buccal mucosa at the implant site.

Secondary outcome measures include 3D hard and soft tissue changes as well as clinical, aesthetic, patient-reported and clinician-reported outcomes.

DETAILED DESCRIPTION:
Patient selection Patients in need of a single implant in the premaxilla (15-25) will be included in this multicenter RCT following screening and after having received written consent.

Sample size calculation A sample size calculation using the Pearson Chi-square test was performed in SAS Power and Sample Size based on a comparison of the proportion on the need for soft tissue augmentation at 5 months following alveolar ridge preservation (ARP) between the control group (ARP + delayed implant placement 'DIP') and test group (ARP + immediate implant placement 'IIP'). The calculation was based on finding a 30% difference between these groups. With alpha set at 0.05 and a power of 0.80, the sample size calculation indicated 28 patients to be included per group. To compensate for drop-outs, 30 patients would be treated with ARP+DIP and 30 would be treated with ARP+IIP.

Clinicians and centers, randomization, allocation concealment and blinding Six experienced clinicians will treat at least 10 patients each. Five clinicians are staff members of the Department of Periodontology and Oral Implantology at UGent - UZ Gent, who also work part-time in different private practices. The final clinician is a professor at the Saint-Luc University Hospital (UCL). The digital workflow, the implant placement protocol, the application of a connective tissue graft (CTG) at 6 months following ARP and the restorative protocol will be thoroughly discussed among the 6 clinicians in a training session before the start of the trial.

During the training session each clinician will receive 5 sealed envelopes internally coded as 'Delayed implant placement' and another 5 as 'immediate implant placement'. Just prior to surgery, a sealed envelope will be randomly selected and opened to reveal the treatment to be conducted. The measuring investigator will not be involved in the treatment of any of the patients and will be blinded to allow unbiased registrations.

Pre-operative digital planning for fabrication of surgical guide A digital workflow will be adopted for every patient for fabrication of a surgical guide prior to tooth extraction. This requires 3D digital implant planning in designated software on the basis of a pre-op low-dose small-field Cone-Beam CT and intra-oral scan. Note that surgical guides for patients in the ARP+DIP group will also be fabricated following patient selection, even though they are only to be used 4 months later.

Control group: ARP+DIP Patients start to take systemic antibiotics (Amoxicilline 1g) and anti-inflammatory medication (Ibuprofen 600 mg) 1h pre-operatively. Following local anesthesia (Septanest special, Septodont, Saint Maur des Fossés, France) and oral disinfection (Corsodyl mouth rinse, GSK, Wavre, Belgium), the failing tooth is extracted without raising a flap. Following socket debridement and rinsing, collagen-enriched DBBM (Bio-Oss Collagen 250 mg, Geistlich Pharma AG, Wolhusen, Switserland) is applied up to the level of the palatal bone crest and slightly condensed. The occlusal aspect is closed with a collagen matrix (Mucograft Seal, Geistlich Pharma AG, Wolhusen, Switserland), which is fixed with single sutures (Seralon 6/0, Serag Weissner, Naila, Germany) to the soft tissues. Post-op instructions include the intake of systemic antibiotics during 4 days (Amoxicilline 1g, two times a day), anti-inflammatory medication as deemed necessary by the patient and oral disinfection twice a day during 1 week. Then, sutures are removed. A removable partial denture as used as provisional tooth replacement when considered needed.

At 4 months, a mucoperiosteal flap is raised, the surgical guide is applied, and the implant is installed according to manufacturer's prescriptions. Then, an implant impression is taken for fabrication of a provisional crown. Prior to wound closure with vertical mattrass sutures (Seralon 6/0, Serag Weissner, Naila, Germany), an appropriate healing abutment is installed. This healing abutment is replaced by the provisional crown two days later.

At 6 months, the need for soft tissue augmentation is assessed by the 5 clinicians who have not been clinically involved. The treating clinician is excluded since he/she cannot be blinded for the treatment group. The need for soft tissue augmentation is assessed on the basis of screenshots from the pre-op CBCT with lip retractors enabling to evaluate buccal bone and soft tissue thickness. Pre-op clinical pictures, clinical pictures at 6 months with the provisional crown in situ and the STL file at 6 months are also offered to the panel in order to assess the loss of buccal convexity.

Soft tissue augmentation is required necessary when at least one of the following criteria are met: thin gingival biotype as defined as < 1mm midfacial soft tissue thickness as assessed on pre-op CBCT with lip retractors, thin buccal bone wall as defined as < 0.5mm as assessed on pre-op CBCT, loss of ideal buccal convexity at 6 months following ARP as assessed on the basis of clinical pictures and STL. Each clinician makes a decision on the need for soft tissue augmentation for 50 out of 60 cases independent from the other clinicians. Soft tissue augmentation is offered to the patient when the majority of the panel is in favor of it.

Soft tissue augmentation is performed using a CTG harvested from the lateral palate using the single incision technique. At the recipient site, a pouch is made in the buccal mucosa and an appropriately sized CTG is pulled in. The CTG is secured into the buccal mucosa with multiple single sutures (Seralon 6/0, Serag Weissner, Naila, Germany) and the provisional crown is re-installed. Sutures are removed after 1 week. The provisional crown is replaced by a permanent crown 3 months later.

Test group: ARP+IIP Patients start to take systemic antibiotics (Amoxicilline 1g) and anti-inflammatory medication (Ibuprofen 600 mg) 1h pre-operatively. Following local anesthesia (Septanest special, Septodont, Saint Maur des Fossés, France) and oral disinfection (Corsodyl mouth rinse, GSK, Wavre, Belgium), the failing tooth is extracted without raising a flap. Following socket debridement and rinsing, the surgical guide is applied, and the implant is installed according to manufacturer's prescriptions. Then, an implant impression is taken for fabrication of a provisional crown. Finally, the gap is filled with collagen-enriched DBBM (Bio-Oss Collagen 250 mg, Geistlich Pharma AG, Wolhusen, Switserland), which is applied up to the level of the free mucosal margin, and an appropriate healing abutment is installed. This healing abutment is replaced by the provisional crown two days later.

At 6 months, the need for soft tissue augmentation is assessed by the 5 clinicians who have not been clinically involved. The treating clinician is excluded since he/she cannot be blinded for the treatment group. The need for soft tissue augmentation is assessed on the basis of screenshots from the pre-op CBCT with lip retractors enabling to evaluate buccal bone and soft tissue thickness. Pre-op clinical pictures, clinical pictures at 6 months with the provisional crown in situ and the STL file at 6 months are also offered to the panel in order to assess the loss of buccal convexity. Each clinician makes a decision on the need for soft tissue augmentation for 50 out of 60 cases independent from the other clinicians. Soft tissue augmentation is offered to the patient when the majority of the panel is in favor of it.

Soft tissue augmentation is performed using a CTG harvested from the lateral palate using the single incision technique. At the recipient site, a pouch is made in the buccal mucosa and an appropriately sized CTG is pulled in. The CTG is secured into the buccal mucosa with multiple single sutures (Seralon 6/0, Serag Weissner, Naila, Germany) and the provisional crown is re-installed. Sutures are removed after 1 week. The provisional crown is replaced by a permanent crown 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* good oral hygiene defined as full-mouth plaque score ≤ 25% (O'Leary et al. 1972)
* presence of a single-rooted tooth in the anterior maxilla (15-25) that needs to be extracted for any reason with at least one neighboring tooth present
* at least 3 mm bone available at the apical or palatal aspect of the alveolus to ensure primary implant stability
* intact or nearly intact buccal bone wall at the time of extraction (max 3 mm bone missing = max 6 mm distance from free gingival margin to buccal bone crest)

Exclusion Criteria:

* systemic diseases
* smoking
* untreated periodontal disease
* untreated caries lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Need for soft tissue augmentation (true or false) as judged by a panel of clinicians | 6 months
  The need for soft tissue augmentation is assessed by the 5 clinicians who have not been clinically involved. The treating clinician is excluded since he/she cannot be blinded for the treatment group. The need for soft tissue augmentation is assessed on the basis of clinical pictures, a CBCT image and STL file.

SECONDARY OUTCOMES:
Clinician-reported outcome measures | per-op
  Ease of implant placement (Visual Analogue Scale). Minimum value = 0 (Very easy) Maximum value = 10 (Very difficult)
Changes in buccal soft tissue profile | pre-op, 6 months, 1 year, 3 years, 5 years
  Volumetric analysis with designated software on the basis of IOS (mm). Change in buccal soft tissue profile and the initial buccal soft tissue profile will be aggregated to calculate relative change in buccal soft tissue profile (=absolute change / initial buccal soft tissue profile, percent)
Vertical change in midfacial soft tissue level | pre-op, 6 months, 1 year, 3 years, 5 years
  Analysed with designated software on the basis of IOS (mm)
Change in width of the alveolar process | pre-op, 1 year, 5 year
  Horizontal measurements with designated software on the basis of CBCT scans (mm)
Change in height of the alveolar process | pre-op, 1 year, 5 year
  vertical measurements with designated software on the basis of CBCT scans (mm)
Change in buccal bone thickness | pre-op, 1 year, 5 year
  Horizontal measurements with designated software on the basis of CBCT scans (mm)
Implant survival | 6 months, 9 months, 1 year, 3 years, 5 years
  presence of the implant
Complication | Up to 5 years
  Any complication
Changes in radiographic outcomes | implant placement, 1 year, 3 years, 5 years
  marginal peri-implant bone level change as assessed by intra-oral radiography (mm)
Aesthetic outcome as assessed by care providers | pre-op, 1 year, 3 years, 5 years
  Pink Aesthetic Score (0-14) = assessment of 7 different parameters (Mesial papilla, distal papilla, tissue contour, gingival level, alveolar process, coloring, texture) which are all rated 0 (worst) - 2 (best)
Aesthetic outcome as assessed by patients | pre-op, 1 year, 3 years, 5 years
  Patients aesthetic satisfaction (Visual Analogue Scale) Minimum value = 0 (Very unsatisfied) Maximum value = 10 (Very satisfied)
Keratinized mucosa width | pre-op, 1 year, 3 years, 5 years
  Vertical measurement performed with a periodontal probe (mm)
Probing pocket depth | pre-op, 1 year, 3 years, 5 years
  Probing depth measured with a periodontal probe (mm)
Bleeding on probing | pre-op, 1 year, 3 years, 5 years
  Bleeding on probing was registered 15 seconds following pocket probing at four sites per implant (mesial, distal, buccal, palatal) using a dichotomous score (0: no bleeding; 1: bleeding). These values were averaged and expressed as a percentage on implant level
Plaque | pre-op, 1 year, 3 years, 5 years
  Plaque was recorded at four sites per implant (mesial, distal, buccal, palatal) using a dichotomous score (0: no visible plaque at the soft tissue margin; 1: visible plaque at the soft tissue margin). These values were averaged and expressed as a percentage on implant level.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Ghent University, Ghent, Oost-Vlaanderen
  - UCL St Luc, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Background] Bittner N, Schulze-Spate U, Silva C, Da Silva JD, Kim DM, Tarnow D, Gil MS, Ishikawa-Nagai S. Changes of the alveolar ridge dimension and gingival recession associated with implant position and tissue phenotype with immediate implant placement: A randomised controlled clinical trial. Int J Oral Implantol (Berl). 2019;12(4):469-480. PMID 31781700
- [Background] Cosyn J, De Bruyn H, Cleymaet R. Soft tissue preservation and pink aesthetics around single immediate implant restorations: a 1-year prospective study. Clin Implant Dent Relat Res. 2013 Dec;15(6):847-57. doi: 10.1111/j.1708-8208.2012.00448.x. Epub 2012 Feb 29. PMID 22376232
- [Background] Cosyn J, Eghbali A, Hermans A, Vervaeke S, De Bruyn H, Cleymaet R. A 5-year prospective study on single immediate implants in the aesthetic zone. J Clin Periodontol. 2016 Aug;43(8):702-9. doi: 10.1111/jcpe.12571. Epub 2016 Jun 13. PMID 27120578
- [Background] Cosyn J, Pollaris L, Van der Linden F, De Bruyn H. Minimally Invasive Single Implant Treatment (M.I.S.I.T.) based on ridge preservation and contour augmentation in patients with a high aesthetic risk profile: one-year results. J Clin Periodontol. 2015 Apr;42(4):398-405. doi: 10.1111/jcpe.12384. Epub 2015 Mar 31. PMID 25728590
- [Background] Kan JY, Rungcharassaeng K, Lozada JL, Zimmerman G. Facial gingival tissue stability following immediate placement and provisionalization of maxillary anterior single implants: a 2- to 8-year follow-up. Int J Oral Maxillofac Implants. 2011 Jan-Feb;26(1):179-87. PMID 21365054
- [Background] Migliorati M, Amorfini L, Signori A, Biavati AS, Benedicenti S. Clinical and Aesthetic Outcome with Post-Extractive Implants with or without Soft Tissue Augmentation: A 2-Year Randomized Clinical Trial. Clin Implant Dent Relat Res. 2015 Oct;17(5):983-95. doi: 10.1111/cid.12194. Epub 2013 Dec 27. PMID 24373419
- [Background] Sanz M, Lindhe J, Alcaraz J, Sanz-Sanchez I, Cecchinato D. The effect of placing a bone replacement graft in the gap at immediately placed implants: a randomized clinical trial. Clin Oral Implants Res. 2017 Aug;28(8):902-910. doi: 10.1111/clr.12896. Epub 2016 Jun 7. PMID 27273298
- [Background] Seyssens L, Eghbali A, Cosyn J. A 10-year prospective study on single immediate implants. J Clin Periodontol. 2020 Oct;47(10):1248-1258. doi: 10.1111/jcpe.13352. Epub 2020 Sep 2. PMID 32748983
- [Background] Yoshino S, Kan JY, Rungcharassaeng K, Roe P, Lozada JL. Effects of connective tissue grafting on the facial gingival level following single immediate implant placement and provisionalization in the esthetic zone: a 1-year randomized controlled prospective study. Int J Oral Maxillofac Implants. 2014 Mar-Apr;29(2):432-40. doi: 10.11607/jomi.3379. PMID 24683571
- [Background] Zuiderveld EG, Meijer HJA, den Hartog L, Vissink A, Raghoebar GM. Effect of connective tissue grafting on peri-implant tissue in single immediate implant sites: A RCT. J Clin Periodontol. 2018 Feb;45(2):253-264. doi: 10.1111/jcpe.12820. Epub 2017 Dec 5. PMID 28941303